CLINICAL TRIAL: NCT03806556
Title: A Pediatric Trial Using Tranexamic Acid in Thrombocytopenia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual rate, strategic reasons
Sponsor: Meghan McCormick (Other)
Responsible Party: Sponsor-Investigator, Meghan McCormick, Principal Investigator, Fellow, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO18100519
Record Dates: First submitted 2019-01-04; First posted 2019-01-16 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Cancer; Thrombocytopenia; Hemostatic Disorder; Coagulation Defect; Acquired
Keywords: tranexamic acid; anti-fibrinolytic agents; chemotherapy-induced thrombocytopenia
MeSH Terms: conditions — Neoplasms; Thrombocytopenia; Hemostatic Disorders | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: This trial is designed as a prospective, randomized, controlled, blinded (patient, caregiver, physician, assessor) trial with two parallel groups and a primary endpoint of feasibility and safety. Randomization will be performed as block randomization with a 1:1 allocation within blocks of size four.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational pharmacy will be notified when patients enroll on trial. When participants meet criteria for randomization, this will be completed by the Investigational Pharmacy. The pharmacy will prepare and distribute to floor nursing staff all doses of tranexamic acid (available in IV form as a colorless liquid) or placebo (as an equal volume of normal saline). Labels will not carry identifiers of which study arm the enrolled patient is on.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Experimental): Doses will be given intravenous (IV). Doses are administered every 8 hours or three times daily (TID) per the discretion of the treating investigator. TXA dose will be 10mg/kg, diluted in normal saline to a total volume of 15 milliliters (mL).
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Doses will be given intravenous (IV). Doses are administered every 8 hours or TID per the discretion of the treating investigator. Normal saline will be administered at a total volume of 15mL.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — IV medication administered after patient meets inclusion/exclusion criteria
  Other Names: TXA
  Arms: Tranexamic Acid
Drug: Normal saline — IV medication administered after patient meets inclusion/exclusion criteria
  Other Names: NS
  Arms: Placebo

SUMMARY:
This study evaluates the use of tranexamic acid (TXA) in addition to standard therapy in children receiving chemotherapy or blood and/or marrow transplantation to decrease the risk of bleeding. Half of participants will receive tranexamic acid and half of participants will receive placebo.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a prospective, randomized, blinded, placebo controlled trial to evaluate the safety and feasibility of the addition of antifibrinolytic therapy with tranexamic acid to the standard care in patients who are thrombocytopenic due to primary bone marrow disorders or chemotherapy, immunotherapy and/or radiation therapy in order to prevent bleeding. The results of this study will change practice by providing evidence as to whether or not TXA is effective and safe treatment when used as an adjunct to platelet transfusion therapy in the thrombocytopenic patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of hematologic malignancy or solid tumor malignancy
* Patients must be undergoing or planned chemotherapy or BMT
* Patients will only be eligible to receive study drug or placebo during inpatient periods
* Patients must be predicted to have thrombocytopenia ≤20,000/microliter (uL) for ≥5 days
* Patient must have a platelet transfusion threshold of ≤30,000/uL
* Patients must be >14 days beyond their last dose of Pegylated(PEG)-Asparaginase or >72 hours beyond their last dose of Erwinia Asparaginase
* Patients must be able to comply with treatment and monitoring

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL)
* History of Immune Thrombocytopenic Purpura (ITP), Thrombotic Thrombocytopenic Purpura (TTP) or Hemolytic Uremic Syndrome (HUS)
* Diagnosis of Disseminated Intravascular Coagulopathy (DIC)
* History of inherited or acquired bleeding disorder AND/OR inherited or acquired prothrombotic disorder
* Patient must not have WHO Grade 2 bleeding or greater within 48 hours prior to enrollment or study drug activation
* Patient must not have received PEG-Asparaginase within the 7 day period prior to enrollment. If given within the 8-14 day period prior to enrollment patients are eligible if prothrombin time (PT), partial thromboplastin time (PTT), international normalized ratio (INR) and fibrinogen are obtained and are within 1.5 times the upper limits of normal.
* Patient must not be receiving tranexamic acid or other anti-fibrinolytic agent or any other agent to promote hemostasis (which includes DDAVP, recombinant Factor VII, Prothrombin Complex Concentrate, Estrogen Derivatives and Progestins)
* Patient must not be receiving therapy with anticoagulation or antiplatelet therapy (which includes heparin infusion, enoxaparin, aspirin. If anticoagulant/antiplatelet therapy is discontinued when platelet count is <50,000/uL patient will be eligible for enrollment)
* Patient must not be receiving platelet growth factors
* Current thromboembolic event
* History of thromboembolic event <6 months prior to enrollment
* Current/prior history of sinusoidal obstruction disease
* Visible hematuria
* Renal dysfunction (as defined by age-specific creatinine values calculated by Schwartz equation) or hemodialysis or anuria (defined as <10 mL urine/hour over 24 hours)
* History of seizures
* Allergy to tranexamic acid
* Pregnancy
* Unwilling to accept blood product transfusions

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan McCormick, MD, Principal Investigator — UPMC Childrens Hospital of Pittsburgh
Locations (1):
- UPMC Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized public data set will be available after publication of primary results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning within 1 year and ending 5 years after trial completion
Access Criteria: Researchers who provide a methodologically sound proposal may request data. Proposals should be directed to meghan.mccormick3@chp.edu. To gain access data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 9.5 [3 to 18] | 11 [3 to 12] | 11 [3 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Diagnosis [Count of Participants; unit: Participants]
  Lymphoid Leukemia | 4 | 0 | 4
  Myeloid Leukemia | 0 | 2 | 2
  Lymphoma | 1 | 1 | 2
  Solid Tumor | 1 | 2 | 3
Type of Therapy [Count of Participants; unit: Participants]
  Chemotherapy | 4 | 2 | 6
  Autologous Hematopoietic Stem Cell Transplant | 1 | 2 | 3
  Allogeneic Hematopoietic Stem Cell Transplant | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Tranexamic Acid in Participants as the Number of Patients With Any Adverse Events and Serious Adverse Events (SAE) as Assessed by CTCAE v4.03
Description: Adverse Events and Serious Adverse Events (SAE) will be collected on subjects throughout their participation in the study and up to 30 days following discontinuation of the study drug, regardless of attribution. Adverse events and serious adverse events will be tabulated by type and grade according to the NCI CTCAE v 4.03.
  The hypothesis is that tranexamic acid can be safely added to standard care regimens in patients with hematologic malignancies or solid tumors during periods of severe thrombocytopenia. Analysis limited to a descriptive assessment of the safety of tranexamic acid in patients with hematologic malignancies or solid tumors by reported adverse events, serious adverse events and death.
Time Frame: From activation of the study drug (maximum 30 days) through 30 days from discontinuation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Grade 3 Adverse Events : Anemia | 4 | 4
  Grade 3 Adverse Events : Anorexia | 0 | 2
  Grade 3 Adverse Events : Bone Pain | 1 | 0
  Grade 3 Adverse Events : Catheter Related Infection | 3 | 1
  Grade 3 Adverse Events : Vomiting | 0 | 2
  Grade 3 Adverse Events : Febrile Neutropenia | 2 | 3
  Grade 3 Adverse Events : Fever | 0 | 1
  Grade 3 Adverse Events : Hypoalbuminemia | 1 | 0
  Grade 3 Adverse Events : Hypotension | 0 | 1
  Grade 3 Adverse Events : Hypoxia | 0 | 1
  Grade 3 Adverse Events : Hypophosphatemia | 0 | 1
  Grade 3 Adverse Events : Rash Maculo-Papular | 0 | 2
  Grade 3 Adverse Events : Nausea | 0 | 1
  Grade 3 Adverse Events : Mucositis Oral | 0 | 1
  Grade 3 Adverse Events : Sinusitis | 0 | 1
  Grade 3 Adverse Events : Skin Infection | 1 | 0
  Grade 3 Adverse Events : White Blood Cell Decreases | 0 | 0
  Grade 3 Adverse Events : Platelet Count Decreased | 0 | 0
  Grade 3 Adverse Events : Blood Bilirubin Increased | 0 | 0
  Grade 4 Adverse Events : Anemia | 0 | 0
  Grade 4 Adverse Events : Anorexia | 0 | 0
  Grade 4 Adverse Events : Bone Pain | 0 | 0
  Grade 4 Adverse Events : Catheter Related Infection | 0 | 0
  Grade 4 Adverse Events : Vomiting | 0 | 0
  Grade 4 Adverse Events : Febrile Neutropenia | 0 | 1
  Grade 4 Adverse Events : Fever | 0 | 0
  Grade 4 Adverse Events : Hypoalbuminemia | 0 | 0
  Grade 4 Adverse Events : Hypotension | 0 | 0
  Grade 4 Adverse Events : Hypoxia | 0 | 0
  Grade 4 Adverse Events : Hypophosphatemia | 0 | 0
  Grade 4 Adverse Events : Rash Maculo-Papular | 0 | 0
  Grade 4 Adverse Events : Nausea | 0 | 0
  Grade 4 Adverse Events : Mucositis Oral | 0 | 0
  Grade 4 Adverse Events : Sinusitis | 0 | 0
  Grade 4 Adverse Events : Skin Infection | 0 | 0
  Grade 4 Adverse Events : White Blood Cell Decreases | 6 | 5
  Grade 4 Adverse Events : Platelet Count Decreased | 6 | 5
  Grade 4 Adverse Events : Blood Bilirubin Increased | 1 | 0

2. Primary Outcome: Feasibility of Tranexamic Acid as an Adjunct to Standard Therapy: Number of Participants Eligible and Recruited
Description: Number of participants eligible for study enrollment and recruited.
  The hypothesis is that tranexamic acid can be safely added to standard care regimens in patients with hematologic malignancies or solid tumors during periods of severe thrombocytopenia. A descriptive assessment of feasibility of recruitment by monitoring number of patients screened, number of patients eligible for enrollment and rate of recruitment (both start-up and ongoing) during study period to be completed by collecting data on the number of patients screened, the number of patients eligible for study inclusion, the number of eligible patients who consent to study inclusion and the number of consented patients activated to the study drug, organized in visual form by CONSORT diagram.
Time Frame: From time of recruitment of the first patient until the last patient is enrolled, up to 16 months in duration
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: All patients assessed for eligibility as defined by diagnosis of hematologic or solid tumor malignancy and anticipated platelet counts ≤20,000/uL for ≥5 days
Arm/Group | Overall Study
Number analyzed (Participants) | 693
Participants
  Assessed for Eligibility | 693
  Screened for Complete Inclusion/Exclusion Criteria | 148
  Eligible for Enrollment | 31
  Consented to Participate | 11

3. Secondary Outcome: World Health Organization (WHO) Bleeding Scale Grade 2 or Higher Bleeding
Description: Proportion of patients with bleeding of WHO grade 2 or above, after activation of study drug. Bleeding graded on a scale ranging from 1 (minor bleeding) through 4 (bleeding that is fatal or life-threatening).
Time Frame: 30 days after activation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 0 | 3

4. Secondary Outcome: Number of Platelet and Red Blood Cell Transfusions
Description: Number of platelet and red blood cell transfusions per patient during the first 30 days post prescription activation of study drug
Time Frame: 30 days after activation of study drug
Measure: Median (Full Range); unit: transfusions
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
transfusions
  Number of platelet transfusions per patient | 1.5 [0 to 2] | 4 [1 to 9]
  Number of pRBC transfusions per patient | 0.5 [0 to 3] | 1 [0 to 2]

5. Secondary Outcome: Number of Days Alive and Without WHO Grade 2 Bleeding or Greater
Description: Number of days alive and without WHO grade 2 bleeding or greater during the first 30 days post activation of study drug. Bleeding graded on a scale ranging from 1 (minor bleeding) through 4 (bleeding that is fatal or life-threatening).
Time Frame: 30 days after activation of study drug
Measure: Mean (Full Range); unit: days
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
days | 5.5 [2 to 8] | 10.4 [1 to 18]

6. Secondary Outcome: The Occurrence of Thromboembolic Adverse Events and Serious Adverse Events
Description: Any venous or arterial thrombosis on standard diagnostic imaging post-randomization
Time Frame: From activation of the study drug (maximum 30 days) through 30 days from discontinuation of study drug
Measure: Number; unit: events
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
events | 0 | 0

7. Secondary Outcome: Bleeding of Any Grade
Description: Proportion of patients with bleeding of any grade as assessed by WHO bleeding score, after activation of study drug
Time Frame: From activation of the study drug (maximum 30 days) through 30 days from discontinuation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 4 | 5

8. Secondary Outcome: Highest Observed Grade of Bleeding (as Measured on WHO Bleeding Scale) During the Study Period
Description: Highest grade of bleeding (as measured on WHO bleeding scale) during study period in each enrolled patient. Bleeding graded on a scale ranging from 1 (minor bleeding) through 4 (bleeding that is fatal or life-threatening).
Time Frame: From activation of the study drug (maximum 30 days) through 30 days from discontinuation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Grade 1 Bleeding | 4 | 2
  Grade 2 Bleeding | 0 | 3
  Grade 3 Bleeding | 0 | 0
  Grade 4 Bleeding | 0 | 0
  Grade 5 Bleeding | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of activation of the study drug up to and including 30 days after the last dose of the study drug, an average of 41 days
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 6/6 | 5/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (N=6) | Placebo (N=5)
White Blood Cell Decreased (Blood and lymphatic system disorders) | 6 | 5 — Grade 4
Platelet Count Decreased (Blood and lymphatic system disorders) | 6 | 5 — Grade 4
Blood Bilirubin Increased (Hepatobiliary disorders) | 1 | 0 — Grade 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 — Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (N=6) | Placebo (N=5)
Anemia (Blood and lymphatic system disorders) | 4 | 4 — Anemia (Grade 3)
Anorexia (Metabolism and nutrition disorders) | 0 | 2 — Anorexia (Grade 3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Bone Pain (Grade 3)
Catheter Related Infection (Infections and infestations) | 3 | 1 — Catheter Related Infection (Grade 3)
Vomiting (Gastrointestinal disorders) | 0 | 2 — Vomiting (Grade 3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 3 — Febrile Neutropenia (Grade 3)
Fever (General disorders) | 0 | 1 — Fever (Grade 3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 — Hypoalbuminemia (Grade 3)
Hypotension (Vascular disorders) | 0 | 1 — Hypotension (Grade 3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Hypoxia (Grade 3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 — Hypophosphatemia (Grade 3)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 — Rash Maculo-papular (Grade 3)
Nausea (Gastrointestinal disorders) | 0 | 1 — Nausea (Grade 3)
Mucositis Oral (Gastrointestinal disorders) | 0 | 1 — Mucositis Oral (Grade 3)
Sinusitis (Infections and infestations) | 0 | 1 — Sinusitis (Grade 3)
Skin Infection (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
The pre-specified analysis described in the study protocol stated the following: "For secondary endpoints, events of WHO Grade 2 or higher bleeding will be compared through the use of odds ratio or T-test statistic of means. The mean number of platelet transfusions will be analyzed using a T-test statistic of means." This analysis was not completed as it would be scientifically inappropriate due to insufficient enrollment. Instead a descriptive analysis was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT03806556/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT03806556/ICF_001.pdf